CLINICAL TRIAL: NCT06716879
Title: A Single-Center, Randomized, Investigator- and Participant-Blind, Placebo-Controlled, Phase 1 Study to Evaluate Safety, Tolerability, and Pharmacokinetics After a Single Dose of Donzakimig in Healthy Chinese and Japanese Participants
Brief Title: A Study to Evaluate Safety, Tolerability, and Pharmacokinetics of a Single Dose of Donzakimig in Healthy Chinese and Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UP0142
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: donzakimig; UCB1381; Phase 1; Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Low Dose of donzakimig in Chinese participants (Experimental): Chinese participants will be randomized to receive a predefined dosage of donzakimig.
  Interventions: Drug: Donzakimig
- High Dose of donzakimig in Chinese participants (Experimental): Chinese participants will be randomized to receive a predefined dosage of donzakimig.
  Interventions: Drug: Donzakimig
- Low Dose of placebo in Chinese participants (Placebo Comparator): Chinese participants will be randomized to receive a predefined dosage of placebo.
  Interventions: Drug: Placebo
- High Dose of placebo in Chinese participants (Placebo Comparator): Chinese participants will be randomized to receive a predefined dosage of placebo.
  Interventions: Drug: Placebo
- Low Dose of donzakimig in Japanese participants (Experimental): Japanese participants will be randomized to receive a predefined dosage of donzakimig.
  Interventions: Drug: Donzakimig
- High Dose of donzakimig in Japanese participants (Experimental): Japanese participants will be randomized to receive a predefined dosage of donzakimig.
  Interventions: Drug: Donzakimig
- Low Dose of placebo in Japanese participants (Placebo Comparator): Japanese participants will be randomized to receive a predefined dosage of placebo.
  Interventions: Drug: Placebo
- High Dose of placebo in Japanese participants (Placebo Comparator): Japanese participants will be randomized to receive a predefined dosage of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donzakimig — Drug: Donzakimig Pharmaceutical form: Subcutaneous solution
  Other Names: UCB1381
  Arms: High Dose of donzakimig in Chinese participants; High Dose of donzakimig in Japanese participants; Low Dose of donzakimig in Chinese participants; Low Dose of donzakimig in Japanese participants
Drug: Placebo — Drug: Placebo Pharmaceutical form: Subcutaneous solution
  Arms: High Dose of placebo in Chinese participants; High Dose of placebo in Japanese participants; Low Dose of placebo in Chinese participants; Low Dose of placebo in Japanese participants

SUMMARY:
The purpose of the study is to investigate the safety, tolerability, and pharmacokinetic parameters of 2 dose strengths of donzakimig, each administered subcutaneously as a single dose, in healthy Chinese and Japanese study participants.

ELIGIBILITY:
Inclusion criteria

* Study participant must be 18 to 55 years of age inclusive at the time of signing the informed consent form (ICF)
* Study participant who is overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac assessment
* Chinese study participant who is of Chinese descent as evidenced in appearance and verbal confirmation of familial heritage and is of Chinese descent with all 4 grandparents, OR Japanese study participant who is of Japanese descent as evidenced in appearance and verbal confirmation of familial heritage and is of Japanese descent with all 4 grandparents
* Study participant has a body mass index within the range of 18 to 30kg/m2 (inclusive)
* Study participant can be male or female

Exclusion criteria

* Study participant has clinically significant multiple or severe drug allergies (including to humanized monoclonal antibodyies (mAbs), intolerance to topical corticosteroids, severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis), known relevant allergy (not including mild seasonal hay fever and/or conjunctivitis or low grade food intolerances), pre-existing history of a relevant allergic condition, or a predisposition for an allergic reaction, as judged by the Investigator
* Study participant has a recent history (within 6 months prior to Screening) or currently active clinically-significant bacterial, fungal, endoparasite (including the presence of ova, cysts, or parasites detected in stool sample provided at Screening), or viral (including hospitalization for coronavirus disease 2019 [COVID-19]) infection, as judged by the Investigator
* Study participant has a history of inflammatory bowel disease (eg, Crohn's disease or ulcerative colitis)
* Study participant has a history of diabetes
* Study participant has received any vaccination within 8 weeks for live vaccines (including attenuated) and 4 weeks for nonlive vaccines prior to the Baseline Visit or is anticipated to do so within 60 days after the dose of IMP
* Study participant has received Bacillus Calmette-Guerin vaccinations within 1 year prior to the Baseline Visit or will receive them within 90 days after the dose of IMP
* Study participant has participated in another study of an IMP or has received any biologic agent within the 30 days prior to Screening (or 5 half-lives, whichever is longer)
* Study participant has had a positive human immunodeficiency virus (HIV) antibody test
* Study participant has the presence of either hepatitis B core antibody or hepatitis B surface antigen at Screening or within 3 months prior to dosing
* Study participant has a positive hepatitis C antibody test result at Screening or within 3 months prior to Screening.
* Study participant has a positive hepatitis C ribonucleic acid (RNA) test result at Screening or within 3 months prior to Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent adverse events (TEAEs) | From Baseline to End of Study visit (up to Day 57)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment emergent adverse events (TEAEs) are adverse events not present prior to the pharmaceutical product administration or an already present event that worsens either in intensity or frequency
Occurrence of serious treatment-emergent adverse events (serious TEAEs) | From Baseline to End of Study visit (up to Day 57)
  A serious treatment-emergent adverse event (serious TEAE) is defined as any untoward medical occurrence that, at any dose:
  Results in death Is life-threatening Requires inpatient hospitalization or prolongation of existing hospitalization Results in persistent disability/incapacity Is a congenital anomaly/birth defect Important medical events
Maximum plasma concentration (Cmax) of donzakimig | Sampling timepoints will be on Day 1 (D1): at predose and 6 hours (h), 24h (D2), 72h (D4), 120h (D6), D8, D15, D22, D36, and D57 after investigational medicinal product (IMP) administration.
  Cmax: Maximum plasma concentration of donzakimig
Area under the plasma concentration-time curve from time 0 to t of donzakimig | Sampling timepoints will be on Day 1 (D1): at predose and 6 hours (h), 24h (D2), 72h (D4), 120h (D6), D8, D15, D22, D36, and D57 after investigational medicinal product (IMP) administration.
  AUC0-t: Area under the plasma concentration-time curve from from 0 to the time (t) of the last quantifiable concentration.
Area under the plasma concentration-time curve from zero to infinity of donzakimig | Sampling timepoints will be on Day 1 (D1): at predose and 6 hours (h), 24h (D2), 72h (D4), 120h (D6), D8, D15, D22, D36, and D57 after investigational medicinal product (IMP) administration.
  AUC: Area under the plasma concentration-time curve from zero to infinity of donzakimig

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 0018445992273
Locations (1):
- UP0142 1, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.